CLINICAL TRIAL: NCT05210335
Title: RISK ANALYSIS AND MANAGEMENT FOR MEDICATION OPTIMIZATION IN THE PREOPERATIVE AND POSTOPERATIVE PERIOD OF CARDIAC SURGICAL PATIENTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Burcu Kelleci Cakir, Lecturer, Hacettepe University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Clinical Pharmacy
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Drug Related Problems; Clinical Pharmacy; Cardiac Surgery; Risk Assesment
Keywords: Drug related problems; Clinical pharmacy; Cardiac surgery; Risk assesment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observational part (No Intervention): This part covers the list for comprehensive medication use at admission, medication reconciliation and medication review at preoperative surgical ward, postoperative intensive care, postoperative surgical ward and discharge made by clinical pharmacist. The identification and classification of drug related problems was made at each ward according to PCNE classification system. The expert panel (2 surgeon, 2 nurse, 1 pharmacist) scored all the drug related problems as a part of the risk analysis model development. Patients quality of life, nutritional status, cognitive functions and frailty status also recorder at admission, discharge and 1 month after surgery.
- Interventional part (Experimental): This part covers the list for comprehensive medication use at admission, medication reconciliation and medication review at preoperative surgical ward, postoperative intensive care, postoperative surgical ward and discharge made by clinical pharmacist. Clinical pharmacist made recommendation about drug related problems regarding solutions, record intervention type and problem status differently from observational part. As a component of the risk analysis model the affect of clinical pharmacist was shown clearly. Patients quality of life, nutritional status, cognitive functions and frailty status also recorder at admission, discharge and 1 month after surgery.
  Interventions: Other: Clinical pharmacist's recommendation to physicians about drug related problems

INTERVENTIONS:
Other: Clinical pharmacist's recommendation to physicians about drug related problems — Clinical pharmacist's recommendation to physicians about drug related problems
  Arms: Interventional part

SUMMARY:
Optimal perioperative and long-term success in cardiac-surgery require precise management of drug treatment. This study was aimed to determine prevalence, types and associated factors of drug related problems (DRPs) at both preoperative and postoperative stages in patients at cardiac-surgery by using risk analysis method.

DETAILED DESCRIPTION:
Cardiac surgery becomes a life-saving option in patients once medical treatments become inadequate. In order to achieve optimal perioperative and long- term success in cardiac surgery, drug treatment should be managed precisely. Patients with cardiovascular diseases are at risk for developing drug related problems (DRPs) due to polypharmacy and having received high-alert medications, such as antiarrhythmics or antithrombotic agents. In addition, type of operation (multiple artery bypass or combined valve procedures), existence of chronic atherosclerotic diseases (such as diabetes mellitus, hypertension), length of stay (LOS) at hospital, frailty, changes in medications for unstable cardiac conditions, incomplete or inadequate history for medication at hospital admission, transition between wards by different healthcare teams and transfer of discrepancies throughout entire perioperative period contributes to increased risk of DRPs in patients at cardiac surgery. It has been shown that over one third of patients suffer from DRPs during hospitalization. Clinical pharmacists are in a position to identify and prevent DRPs, therefore can help to provide optimal pharmaceutical treatment by performing medication reconciliation, improving patient compliance, monitoring of laboratory values and conducting patient education for surgical patients.However, there is limited information about prevalence and risk factors of DRPs in patients at cardiac surgery, in particular with perioperative stages. Majority of studies regarding DRPs have been conducted in specific populations such as elderly, pediatrics or in general medicine. Therefore this study was aimed to determine prevalence, types and associated factors of drug related problems (DRPs) at both preoperative and postoperative stages in patients at cardiac-surgery by using risk analysis method.

ELIGIBILITY:
Inclusion Criteria:

* Patients are aged 18 years or older
* admitted to the hospital for a planned elective cardiac surgery during the study period were considered eligible.

Exclusion Criteria:

* Patients who refused to participate,
* transferred from different wards
* have urgent surgery planned were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Obtaining drug related problems preoperative and postoperative periods | 6 months (1 November 2019-30 March 2020)
  Obtaining valid drug related problems and their characteristic is the primary outcome as a part of the risk analysis.
Building risk analysis model | 3 months (30 March 2020-30 June 2020)
  In line with the valid drug related problems expert panel build the model
Obtaining clinical pharmacist affect | 6 months (1 August 2020- 30 January 2021)
  Obtaining clinical pharmacist affect as a part of the risk analysis model

SECONDARY OUTCOMES:
Obtaining clinical pharmacist intervention on other factors | 6 months (1 August 2020- 30 January 2021)
  the affect of this model on quality of life, nutritional status, fraility status, hospital mortality rate, length of hospital stay, lenght of intensive care unit stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Pharmacy Department of Clinical Pharmacy, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
This will evaluate upon request